CLINICAL TRIAL: NCT03463122
Title: Virtual Reality Based Visual Perception Evaluation and Rehabilitation-pilot Study
Brief Title: Head Mount Display-based Virtual Reality Rehabilitation of Hemispatial Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Collaborators: Hanyang University (Other)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager of Department of Neurorehabilitation, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2014-04-022
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Neglect, Hemispatial
Keywords: stroke; neglect; virtual reality; head mount display; rehabilitation
MeSH Terms: conditions — Stroke; Perceptual Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training first (Other): This group completed 20 sessions of a field of regard-focused visual exploration therapy program using an head mount display (five daily sessions per week over a period of four weeks) in addition to conventional therapy followed by four weeks of conventional therapy
  Interventions: Device: field of regard-focused visual exploration therapy; Other: conventional therapy
- Waiting first (Other): This group completed four weeks of conventional therapy followed by 20 sessions of a field of regard-focused visual exploration therapy program using an head mount display (five daily sessions per week over a period of four weeks) in addition to conventional therapy.
  Interventions: Device: field of regard-focused visual exploration therapy; Other: conventional therapy

INTERVENTIONS:
Device: field of regard-focused visual exploration therapy — field of regard-focused visual exploration therapy in addition to conventional therapy
  Other Names: head mount display
Other: conventional therapy — conventional therapy for stroke rehabilitation

SUMMARY:
Head-mounted display based virtual reality rehabilitation for hemispatial neglect.

DETAILED DESCRIPTION:
The investigators examine about the efficacy of field-of-regard-focused visual exploration therapy implemented using a head-mounted display virtual reality system for hemispatial neglect rehabilitation following stroke.

ELIGIBILITY:
Inclusion Criteria:

* presence of left hemispatial neglect as demonstrated by a score above the cut-off on the line bisection test or star cancellation test of the Behavioral Inattention Test, or mild-to-moderate neglect-related functional impairment defined by a score of 1-20 points on the Catherine Bergego Scale
* age 19 to 65 years
* first-time right hemispheric ischemic or haemorrhagic stroke as evidenced by brain imaging and medical records
* a score >25 on the Mini-Mental State Examination

Exclusion Criteria:

* presence of oculomotor palsies or visual defects as assessed via standard neurological examination
* orthopaedic disorders affecting neck movement
* inability to maintain a seated position.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Field of regard-response time | Baseline, 4 weeks from baseline, 8 weeks from baseline
  time interval between target onset and response with field of regard setting
Change in Field of regard-success rate | Baseline, 4 weeks from baseline, 8 weeks from baseline
  percentage of correct responses (clicking the left or right mouse button in response to a blue or red target, respectively) with field of regard setting
Change in Field of regard-head movement | Baseline, 4 weeks from baseline, 8 weeks from baseline
  sum of all quantified head-rotations with field of regard setting

SECONDARY OUTCOMES:
Field of view-response time | Baseline, 4 weeks from baseline, 8 weeks from baseline
  time interval between target onset and response with field of view setting
Field of view-success rate | Baseline, 4 weeks from baseline, 8 weeks from baseline
  percentage of correct responses (clicking the left or right mouse button in response to a blue or red target, respectively) with field of view setting
Line bisection test | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Participants were asked to bisect the given lines by marking the centre of each line using their preferred or unaffected hand
Star cancellation test | Baseline, 4 weeks from baseline, 8 weeks from baseline
  The experimenter crossed out the two small, central stars of the sheet as an example, following which participants were asked to mark the remaining small stars.
Catherine Bergego Scale | Baseline, 4 weeks from baseline, 8 weeks from baseline
  a standardised checklist designed to detect the degree of neglect during everyday life via direct observation of functioning during ten tasks

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, Principal Investigator — National Rehabilitation Center of Korea
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

REFERENCES:
- [Derived] Shin JH, Kim M, Lee JY, Kim MY, Jeon YJ, Kim K. Feasibility of hemispatial neglect rehabilitation with virtual reality-based visual exploration therapy among patients with stroke: randomised controlled trial. Front Neurosci. 2023 Apr 20;17:1142663. doi: 10.3389/fnins.2023.1142663. eCollection 2023. PMID 37152602
- [Derived] Kim TL, Kim K, Choi C, Lee JY, Shin JH. FOPR test: a virtual reality-based technique to assess field of perception and field of regard in hemispatial neglect. J Neuroeng Rehabil. 2021 Feb 18;18(1):39. doi: 10.1186/s12984-021-00835-1. PMID 33602254